CLINICAL TRIAL: NCT05414760
Title: Evaluation of Adhesions Formation Using Conventional Third Generation Endometrial Ablation With and Without Postoperative Application of an Intrauterine Adhesion Barrier Film
Brief Title: Evaluate Formation of IUAs After Third-generation Endometrial Ablation, With and Without Intrauterine Adhesion Barrier
Acronym: CLEAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Remko P. Bosgraaf (Other)
Responsible Party: Sponsor-Investigator, Remko P. Bosgraaf, Principal Investigator, Catharina Ziekenhuis Eindhoven
Organization: Catharina Ziekenhuis Eindhoven (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CLEAN
Record Dates: First submitted 2022-05-29; First posted 2022-06-10 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Asherman Syndrome; Intrauterine Adhesion
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Womed Leaf group (Active Comparator): Womed Leaf is inserted immediately after completion of the endometrial ablation.
  Interventions: Device: Womed Leaf
- No adhesion prevention group (No Intervention): Standard of care: no IUA prevention, no placebo after ablation

INTERVENTIONS:
Device: Womed Leaf — Womed Leaf™ is a sterile, degradable film of poly(D,L-lactide) (PLA) and poly(ethylene oxide) (PEO). PEO is a biocompatible polymer with anti-adhesion and swelling properties. It is polymerized with hydrophobic PLA to form a degradable film. Womed Leaf™ is inserted in the uterine cavity by a gynaecologist surgeon with a 5 mm diameter flexible inserter. Once released, the film unfolds and grows into the uterine cavity to create a mechanical barrier and keep the uterine walls separated for approximately one week. It is then degraded and discharged naturally through the cervix.
  Arms: Womed Leaf group

SUMMARY:
Evaluate the formation of adhesions after third-generation endometrial ablation, with and without the intrauterine adhesion barrier.

DETAILED DESCRIPTION:
The application of endometrial ablation (EA) has significantly increased in the past 10 years. It is an effective treatment for heavy menstrual bleeding with functional aetiology. However, the risk of post-ablative intracavitary scarring after EA is significant and can lead to long term complications, and the possible delay in diagnosing endometrial cancer. CLEAN is a prospective, multi-center, randomized, controlled, two arm pilot clinical trial. The objective is to compare the formation of adhesions after third-generation endometrial ablation, with and without the intrauterine adhesion barrier.

The study will be performed on women with heavy menstrual bleeding (menorrhagia) scheduled for thermal endometrial ablation with Novasure system (Hologic) A follow-up diagnostic hysteroscopy will be performed 4-8 weeks after the ablation procedure to determine the presence and severity of IUAs according to the American Fertility Society.

ELIGIBILITY:
Inclusion Criteria:

* Patient with refractory heavy menstrual bleeding scheduled for endometrial ablation with Novasure system
* Women 30 years old or older;
* Subjects who are willing to provide a written informed consent as approved by the applicable Ethics Committee / IRB prior to participating in this clinical investigation.
* Subjects who can comply with the study follow-up and other study requirements.

Exclusion Criteria:

* Cavity length <4 or >8
* Perforation during ablation procedure
* Previous adhesiolysis procedure or diagnosis of Asherman's disease.
* Abnormal uterine cavity at the time of ablation according to ESHRE classification I to V such as unicornis, bicornis, septate, duplex
* History of cervical or endometrial cancer
* Active pelvic infection or history of pelvic peritonitis
* Known contraindication or hypersensitivity to Womed Leaf component
* Current participation in another clinical investigation that has not yet received the primary endpoint
* Any other condition that makes participation in the study contrary to the patient's best interests.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Efficacy endpoint: AFS scale; a discrete number | 4-8 weeks after surgery
  Focused on the intrauterine adhesion formation following Novasure (i.e. considering only extent of cavity involved and type of adhesions) Extent of IUA => 1 = less than 1/3 of the cavity involved and 4 = more than 2/3.
  Type of IUA => 1 = filmy and 4 = dense. Sum: 1 = very light adhesions and 12 = extremely severe adhesions obstructing the whole cavity.
Safety endpoint 1.1: Assessment of cavity findings | 4-8 weeks after surgery
  Ability to perform a biopsy anywhere within the uterine cavity
Safety endpoint 1.2: Assessment of cavity findings | 4-8 weeks after surgery
  Ability to adequately visualise the endometrium to evaluate for pathologic change
Safety endpoint 1.3: Assessment of cavity findings | 4-8 weeks after surgery
  Qualitative description of the endometrial cavity (i.e. presence of viable endometrium vs cicatricial/fibrotic tissue…)
Serious adverse events | 3 months after surgery
  Number of Serious Adverse Events and Serious Device-related Adverse Events such as postablation syndrome.

SECONDARY OUTCOMES:
Each component of AFS score at second look hysteroscopy | 4-8 weeks after surgery
  Extent of IUA => 1 = less than 1/3 of the cavity involved and 4 = more than 2/3.
  Type of IUA => 1 = filmy and 4 = dense.
Binary rate of intrauterine adhesions on hysteroscopy | 4-8 weeks after surgery
  Yes/ No intrauterine adhesions are present
Change in menstrual bleeding | 3 months after surgery
  Change in menstrual bleeding using Pictorial Blood Loss Assessment Chart
Level of dysmenorrhea | Before surgery and after 3 months
  Painful cramping associated with menstruation; 0 = no symptoms and 5 = very severe symptoms
Level of patient satisfaction on ablation procedure | Immediately after the surgery
  On a scale from 0 to 5 from the worst to the best health care possible; 0 = worst health care possible and 5 = best health care possible
Number of patients complaints | 3 months after surgery
  Number of patient complaints (i.e. complaints related to discharge or dyspareunia)
Number of subjects for whom a second ablation is possible | 4-8 weeks after surgery
  For each subject, the second look evaluator will assess whether it is possible to perform a second ablation if needed.

CONTACTS AND LOCATIONS:
Overall Officials: Remko Bosgraaf, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (2):
- Netherlands (2):
  - Catharina Hospital, Eindhoven
  - St. Jans Gasthuis, Weert

IPD SHARING:
Plan to Share IPD: Yes
The anonymized data will become available and reusable for other researchers upon reasonable request according to GCP and FAIR principles. All research data will be handled confidentially in accordance with legislation and conditions imposed by Autoriteit Persoonsgegevens.
  Individual participant data that underlie the result that will be reported in an article and study protocol may be made available to researchers who provide a methodologically sound proposal, immediately after article publication and during 5 years
Supporting Information: Study Protocol
Time Frame: Immediately after article publication and during 5 years
Access Criteria: Researchers who provide a methodologically sound proposal